CLINICAL TRIAL: NCT03868384
Title: Evaluation of Home Blood Pressure Measurement for the Management of Hypertension in Treated Hypertensive Patients
Brief Title: The Effect of Home Blood Pressure Measurement on the Management of Hypertension
Status: Active, not recruiting | Type: Observational
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Moo-Yong Rhee, Professor, DongGuk University
Other Study IDs: DUMC-C1801
Record Dates: First submitted 2019-02-22; First posted 2019-03-11 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Hypertension; Blood Pressure; Home Blood Pressure Measurement; Ambulatory Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Home blood pressure measurement has been reported to be associated with better clinic blood pressure and daytime blood pressure control. However, no study has evaluated the association between home blood pressure measurement and control of 24-hour ambulatory blood pressure in real world practice.

The purpose of the present study is to investigate the effect of home blood pressure measurement on the control of ambulatory blood pressure in the real world.

The detailed purposes of the present study are (1) to investigate the effects of home blood pressure measurement on the appropriate control of 24-hour ambulatory blood pressure in hypertensive patients treated with antihypertensive drug, (2) to evaluate the effect of home blood pressure measurement on the occurrence of cardiovascular events and target organ damage, (3) to investigate the status and appropriateness of home blood pressure measurement in the real world, and (4) to investigate factors of home blood pressure measurement methods affecting the treatment of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension and taking antihypertensive drugs more than 1 year

Exclusion Criteria:

* Secondary hypertension
* Hypertensive emergency and urgency
* Severe heart failure (NYHA III and IV)
* Angina with 6 months
* Myocardial infarction within 6 months
* Peripheral artery disease within 6 months
* Significant arrhythmia (i.e. ventricular tachycardia and fibrillation, atrial fibrillation, atrial flutter)
* Pregnancy
* Night labor, shift worker
* Those who are currently participating in other clinical studies
* Those who have taken other clinical trial drugs within the past month
* According to the opinion of the researcher, those who have or may have a disease that may interfere with the completion of the study
* History of drug or alcohol dependence within 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypertension who were taking antihypertensive drugs for more than 1 year for treatment of hypertension are recruited through advertising in Goyang City where the hospital is located and Paju City near to the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 701 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference of 24-hour blood pressure control rate | at baseline and 3 years of follow up
  difference of 24-hour blood pressure control rate between patients who measure and do not measure home blood pressure

SECONDARY OUTCOMES:
Difference of daytime blood pressure control rate | at baseline and 3 years of follow up
  Difference of daytime blood pressure control rate between patients who measure and do not measure home blood pressure
Difference of office blood pressure control rate | at baseline and 3 years of follow up
  Difference of office blood pressure control rate between patients who measure and do not measure home blood pressure
Difference of systolic and diastolic blood pressure (office, 24-hour, daytime, nighttime) | at baseline and 3 years of follow up
  Difference of systolic and diastolic blood pressure (office, 24-hour, daytime, nighttime) between patients who measure and do not measure home blood pressure
Rate of home blood pressure measurement | at baseline and 3 years of follow up
  Rate of home blood pressure measurement in study population
Reflection of home blood pressure | at baseline and 3 years of follow up
  Rate of reflecting home blood pressure in the treatment of hypertension at office
cardiovascular disease prevalence and target organ damage | at baseline and 3 years of follow up
  Difference of cardiovascular disease prevalence and target organ damage between patient who do or do not measure home blood pressure
  * Composites of cardiovascular disease: number of participants with non-fatal myocardial infarction, angina pectoris, revascularization of arteries, stroke, transient ischemic attack, atrial fibrillation, heart failure hospitalization, progression to end-stage renal failure or elevation of creatinine more than 2-fold, other undefined cardiovascular events at the discretion of the investigator
  * Target organ damage: left ventricular hypertrophy by electrocardiography, brachial-ankle pulse wave velocity, microalbuminuria
Changes of home blood pressure measurement rate | from baseline to 3 years of follow up
  Changes of home blood pressure measurement rate in study population after 3 year of follow up from baseline
Cardiovascular disease events and target organ damage | during 3 years of follow up from baseline measurement
  Difference of occurrence of cardiovascular disease events and target organ damage between patient who measure and do not measure home blood pressure
  * Composites of cardiovascular disease events: number of participants with first occurrence of non-fatal myocardial infarction, angina pectoris, revascularization of arteries, stroke, transient ischemic attack, atrial fibrillation, heart failure hospitalization, progression to end-stage renal failure or elevation of creatinine more than 2-fold, other undefined cardiovascular events at the discretion of the investigator
  * Target organ damage: left ventricular hypertrophy by electrocardiography, brachial-ankle pulse wave velocity, microalbuminuria from enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
In order to share the IPD, the informed consent from the research participants is required un the Korean law, and the investigators did not get the consent to share at the beginning of this study.

REFERENCES:
- [Derived] Rhee MY, Munakata M, Nah DY, Kim JS, Kim HY. Home blood pressure measurement for hypertension management in the real world: Do not just measure, but share with your physician. Front Cardiovasc Med. 2023 Jan 18;10:1103216. doi: 10.3389/fcvm.2023.1103216. eCollection 2023. PMID 36742078